CLINICAL TRIAL: NCT03060213
Title: Fun For Wellness Online Intervention to Promote Multidimensional Well-Being: A Randomized Controlled Trial in a Community-Based Patient Sample
Brief Title: Fun For Wellness: Online Well-Being Promotion Intervention in a Patient Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Isaac Prilleltensky, Dean of the School of Education and Human Development; Professor; Vice Provost for Institutional Culture, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170001
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Health Promotion
Keywords: Well-Being; e-Health; Randomized Controlled Trial; Self-Efficacy; Interpersonal well-being; Community well-being; Occupational well-being; Physical well-being; Psychological well-being; Economic well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Health

STUDY DESIGN:
Intervention Model Description: The intervention group will be compared to a usual care (UC) control group on outcomes of overall subjective well-being, domain-specific well-being, health-related quality of life, and well-being self-efficacy. The intervention group will participate in online activities for 30 days while UC control group participants will be asked to conduct their lives as usual for the same 30 day period. Both groups will complete assessments during this time period. The UC group will be given access to the intervention for 30 days after all study participants have completed the three survey battery administrations.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants who have completed the full online T1 battery will be randomly assigned in real-time by the computer to either the intervention condition or the UC control condition. Randomization, group assignment, and assessments will be conducted solely by the computer program, so researchers will be blind to participant randomization, group assignment, and participant group identity during assessment times. With regard to group size and power, experience from our prior efficacy study of FFW indicates that for the current study, the computer program will use a 2:1 randomization algorithm so that there are twice as many FFW intervention participants as UC control participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fun For Wellness (FFW) (Experimental): Intervention participants will: 1) watch original videos with vignettes performed by professional actors; 2) read and/or watch mini-lectures that teach skills for behavior change; 3) engage in self-reflection exercises, 4) play original interactive games related to vignettes and mini-lectures; 5) interact with other FFW users via chat room functions and; 6) watch funny narrated video clips about well-being.
  Interventions: Behavioral: Fun For Wellness (FFW)
- Usual Care (UC) (No Intervention): The Usual Care (UC) group will conduct their lives as usual during the 30 day intervention period.

INTERVENTIONS:
Behavioral: Fun For Wellness (FFW) — FFW consists of videos, games, and content teaching 14 skills to support seven drivers of change that promote well-being in I COPPE domains. The drivers form the acronym BET I CAN, which stands for: Behaviors, Emotions, Thoughts, Interactions, Context, Awareness, and Next Steps. B teaches basics of habit formation, including antecedents, behaviors, and consequences and techniques like goal setting, behavior tracking and rewards. E teaches how to build positive emotions and cope with negative ones. T teaches lessons from cognitive behavioral therapy. I builds communication skills such as empathy, listening and assertiveness. C teaches how to create healthier environmental contexts. A aims to increase insight. N emphasizes the need to make plans and anticipate barriers.
  Arms: Fun For Wellness (FFW)

SUMMARY:
Subjective well-being refers to people's level of satisfaction with life as a whole and with multiple dimensions within it. Interventions that promote subjective well-being are important because there is evidence that physical health, mental health, substance use and health care costs may be related to subjective well-being. This randomized controlled trial will evaluate an online intervention, named Fun For Wellness (FFW), designed to promote well-being skills and self-efficacy in six domains of life: interpersonal, community, occupational, physical, psychological, and economic (I COPPE). The Usual Care (UC) control group will be wait-listed. Five hundred (500) community-based adult patient participants will be enrolled. We hypothesize that compared to the UC group, intervention group participants will show greater improvement in their overall subjective well-being, domain-specific well-being, health-related quality of life, and well-being self-efficacy.

DETAILED DESCRIPTION:
Subjective well-being is a positive state affairs in six domains of life: interpersonal, community, occupational, physical, psychological, and economic (I COPPE). The purpose of the study is to evaluate the effectiveness, feasibility, and acceptability of an online intervention named Fun For Wellness (FFW), designed to promote skills and self-efficacy in the multidimensional I COPPE domains of life.

In designing the program we considered the pressing societal need to promote universal health and well-being and prevent stress, illness and disease. Preventable conditions related to lifestyle such as obesity and stress afflict millions of people. Therefore, we saw a need to develop a universal tool for the adult population who would be comfortable with the online platform of FFW. Universal programs have been shown to be effective, for example, in reducing mental health problems in college students.

While face-to-face interventions are effective in preventing serious conditions, they are very labor intensive and limited in reach. The ability to prevent adverse conditions and to enhance healthy behaviors through online interventions creates several opportunities: accessibility, scalability, interactivity, affordability, and fidelity of implementation. A randomized controlled trial of the FFW intervention in an employee sample, found initial evidence for the effectiveness of the FFW intervention. Participants who complied with the FFW intervention had significantly higher subjective well-being, as compared to compliers in the Usual Care group, in multiple I COPPE domains.

For the current study, well-being and self-efficacy measures will be administered at baseline (T1), 30 days-post baseline (T2) and 60 days -post baseline (T3). A maximum of 500 patients will be enrolled. Recruitment will take place on-site through IRB approved study flyers at a community medical center. All other study activities will take place entirely online at a secure website.

Hypothesis 1: Outcome effects: The online well-being program will be more effective than the usual care condition in improving: 1) overall well-being 2) domain well-being, and 3) health related quality of life (HRQOL) over time.

Hypothesis 2: Self-efficacy effect: The online well-being program will be more effective than the usual care condition in improving I COPPE well-being self-efficacy.

Hypothesis 3: Mediating effect: The effect of the online well-being program on- 1) overall well-being, 2) domain well-being and, 3) health related quality of life will be partially mediated by improvements in I COPPE well-being self-efficacy over time.

ELIGIBILITY:
Inclusion Criteria:

* Individual is at least 18 years old
* Individual is a current patient at University of Miami's UHealth Lennar Medical Center
* Individual is not now, nor has ever participated in activities of the Fun For Wellness online program

Exclusion Criteria:

* Individual less than 18 years old
* Individuals who are not current a patient at University of Miami's UHealth Lennar Medical Center
* Individual is now, or has ever participated in activities of the Fun For Wellness online program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Change in overall well-being I COPPE Scale scores between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The primary objective of this study is to determine if FFW improves well-being as measured by change in I COPPE Scale domain scores after 60 days compared to usual care for patient well-being at the University of Miami's UHealth Lennar Medical Center. The investigators will assess the efficacy of FFW on I COPPE overall well-being as measured by the I COPPE Scale overall well-being score.
Change in interpersonal well-being I COPPE Scale score between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The investigators will assess the efficacy of FFW on improving interpersonal well-being as measured by the I COPPE Scale interpersonal well-being score
Change in community well-being I COPPE Scale score between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The investigators will assess the efficacy of FFW on improving community well-being as measured by the I COPPE Scale community well-being score.
Change in occupational well-being I COPPE Scale score between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The investigators will assess the efficacy of FFW on improving occupational well-being as measured by the I COPPE Scale occupational well-being score.
Change in physical well-being I COPPE Scale score between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The investigators will assess the efficacy of FFW on improving physical well-being as measured by the I COPPE Scale physical well-being score.
Change in psychological well-being I COPPE Scale score between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The investigators will assess the efficacy of FFW on improving psychological well-being as measured by the I COPPE Scale psychological well-being score.
Change in economic well-being I COPPE Scale score between baseline and time 3. | baseline (time 1), 30 days (time 2), and 60 days (time 3)
  The investigators will assess the efficacy of FFW on improving economic well-being as measured by the I COPPE Scale economic well-being score.

SECONDARY OUTCOMES:
Change in health-related quality of life (HRQOL)-physical component score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving HRQOL as measured by the SF-36v2 Health Survey physical component (PC) score.
Change in self-efficacy in well-being (SEWB) overall domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB-overall as measured by the Self-Efficacy in Well-Being Domains Scale overall well-being domain score.
Change in self-efficacy in well-being (SEWB) interpersonal domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB-interpersonal as measured by the Self-Efficacy in Well-Being Domains Scale interpersonal well-being domain score.
Change in self-efficacy in well-being (SEWB) community domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB-community as measured by the Self-Efficacy in Well-Being Domains Scale community well-being domain score.
Change in self-efficacy in well-being (SEWB) occupational domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB-occupational as measured by the Self-Efficacy in Well-Being Domains Scale occupational well-being domain score.
Change in self-efficacy in well-being (SEWB) physical domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB- physical as measured by the Self-Efficacy in Well-Being Domains Scale physical well-being domain score.
Change in self-efficacy in well-being (SEWB) psychological domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB- psychological as measured by the Self-Efficacy in Well-Being Domains Scale psychological well-being domain score.
Change in self-efficacy in well-being (SEWB) economic domain score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving SEWB- economic as measured by the Self-Efficacy in Well-Being Domains Scale economic well-being domain score.
Change in self-efficacy in well-being domains (SEWB) overall score between baseline and time 3 will mediate the relationship between the effect of FFW and change in I COPPE overall well-being scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on overall well-being will be partially mediated by improvements in SEWB-overall over time.
Change in self-efficacy in well-being domains (SEWB) interpersonal score between baseline and time 3 will mediate the relationship between the effect of FFW and change in I COPPE interpersonal well-being scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW on interpersonal well-being will be partially mediated by improvements in SEWB-interpersonal over time.
Change in self-efficacy in well-being domains (SEWB) community score between baseline and time 3 will mediate the relationship between the effect of FFW and change in I COPPE community well-being scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW on community well-being will be partially mediated by improvements in SEWB-community over time.
Change in self-efficacy in well-being domains (SEWB) occupational score between baseline and time 3 will mediate the relationship between the effect of FFW and change in I COPPE occupational well-being scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW on occupational well-being will be partially mediated by improvements in SEWB- occupational over time.
Change in self-efficacy in well-being domains (SEWB) physical score between baseline and time 3 will mediate the relationship between the effect of FFW and change in I COPPE physical well-being scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW on physical well-being will be partially mediated by improvements in SEWB- physical over time.
Change in self-efficacy in well-being domains (SEWB) economic score between baseline and time 3 will mediate the relationship between the effect of FFW and change in I COPPE economic well-being scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW on economic well-being will be partially mediated by improvements in SEWB- economic over time.
Change in self-efficacy in well-being domains (SEWB) overall score between baseline and time 3 will mediate the relationship between the effect of FFW and change on Health Related Quality Of Life (HRQOL) physical (PC) score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB-overall over time.
Change in self-efficacy in well-being domains (SEWB) interpersonal score between baseline and time 3 will mediate the relationship between the effect of FFW and change on HRQOL physical component (PC) scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB-interpersonal over time.
Change in self-efficacy in well-being domains (SEWB) community score between baseline and time 3 will mediate the relationship between the effect of FFW and change on HRQOL physical component (PC) scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB-community over time.
Change in self-efficacy in well-being domains (SEWB) occupational score between baseline and time 3 will mediate the relationship between the effect of FFW and change on HRQOL physical component (PC) scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB-occupational over time.
Change in self-efficacy in well-being domains (SEWB) physical score between baseline and time 3 will mediate the relationship between the effect of FFW and change on HRQOL physical component (PC) scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB- physical over time.
Change in self-efficacy in well-being domains (SEWB) psychological score between baseline and time 3 will mediate the relationship between the effect of FFW and change on HRQOL physical component (PC) scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB- psychological over time.
Change in self-efficacy in well-being domains (SEWB) economic score between baseline and time 3 will mediate the relationship between the effect of FFW and change on HRQOL physical component (PC) scores between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess if the effect of FFW and change on HRQOL-PC will be partially mediated by improvements in SEWB-economic over time.

OTHER OUTCOMES:
Change in I COPPE actions total score between baseline and time 3. | baseline, 30 days, and 60 days
  The investigators will assess the efficacy of FFW on improving I COPPE actions as measured by the I COPPE Actions Scale total score.
Strength of the relationship between self-efficacy to comply scores and complier average causal effect (CACE) values over time. | baseline, 30 days, and 60 days
  The investigators will assess the predictive effect of a participant's self-efficacy to comply with the FFW intervention as measured by the Self-Efficacy to Comply Measure score and CACE coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Prilleltensky, Ph.D., Principal Investigator — Dean, School of Education and Human Development; Professor; Vice Provost, Office of Institutional Culture
Locations (1):
- UHealth Lennar Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No